CLINICAL TRIAL: NCT02123667
Title: AssessmenT of smalL Airways involvemeNT In aSthma (ATLANTIS); Multinational, Multicentre, Non-pharmacological Intervention, Cross-sectional and Longitudinal Study.
Brief Title: AssessmenT of smalL Airways involvemeNT In aSthma (ATLANTIS)
Acronym: ATLANTIS
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CCD-01535AC1-01; CCD-01535AC1-01 (Other: Chiesi Farmaceutici)
Record Dates: First submitted 2014-04-24; First posted 2014-04-25 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional bronchoscopy with endobronchial and trans-bronchial biopsy will be applicable in selected sites only in EU and US. Total number of inflammatory cells and quantification of specific cells including eosinophils, T cells and macrophages will be performed. Gene expression profiles (including RNA) will be performed at a later date for future analysis on the pathobiology of asthma which will be defined in future specific protocols
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthmatic patients: asthmatic patients 18 to 65
- Healthy volunteers: Volunteers 18 to 65

SUMMARY:
Multinational, multicentre, non-pharmacological intervention, cross-sectional and longitudinal study.

DETAILED DESCRIPTION:
Large non pharmacological studies on Small Airways Disease

ELIGIBILITY:
Asthmatic patient inclusion criteria

1. Male or female patients aged ≥ 18 and ≤ 65 years, who have signed an Informed Consent form
2. Clinical diagnosis of asthma f

   1. Positive response to methacholine challenge test
   2. Positive response to a reversibility test or
   3. Peak Flow variability (i.e. highest - lowest PEF over the day/mean value of the two, × 100) > 20% or
   4. Documented response (defined as ΔFEV1 ≥ 12% and ≥ 200 mL) after a cycle (e.g., 4 weeks) of regular maintenance anti-asthma treatment.
3. Patients with stable asthma.
4. Current smoker, ex-smoker or lifelong non-smoker Healthy subject inclusion criteria

1. Male or female patients aged ≥ 18 and ≤ 65 years 2. No clinical history of asthma or COPD 3. Current smoker, ex-smoker or lifelong non-smokers 4. Normal spirometry 5. Normal airways responsiveness Asthmatic patient exclusion criteria

1. Cigarette smoking > 10 packyears
2. diagnosis of COPD
3. Asthma exacerbation in the 8 weeks prior to baseline visit
4. Clinical or functional uncontrolled respiratory, haematological, immunologic, renal, neurologic, hepatic, endocrinal or other disease, or any condition that might compromise the results or interpretation of the study.
5. Pregnant or lactating women
6. Participation in an interventional clinical trial <12 weeks preceding baseline visit
7. Inability to comply with study procedures.
8. Alcohol or drug abuse. Healthy subject exclusion criteria

1. Cigarette smoking history > 10 packyears 2. Diagnosed upper and/or lower respiratory disease(s). 3. Clinical or functional uncontrolled haematological, immunologic, renal, neurologic, hepatic, endocrinal or other disease, or any condition that mightp compromise the results or interpretation of the study.

4. Pregnant or lactating women 5. Participation in an interventional clinical trial <12 weeks preceding baseline visit 6. Inability to comply with study procedures. 7. Alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 900 subjects divided into 800 asthmatic patients and 100 healthy controls will be included. Recruitment will be balanced, at the extent possible, in order to achieve at least > 150 patients each for steps 1 - 4 and > 50 patients for step 5 as indicated in the international guidelines (GINA 2012) on the basis of their previous therapy. The 150 healthy controls will be recruited on the basis of absence of respiratory symptoms, airway obstruction and hyper responsiveness.
Sampling Method: Probability Sample
Enrollment: 872 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-03-04 (Actual); Study Completion 2017-03-04 (Actual)

PRIMARY OUTCOMES:
To determine the role of small airways abnormalities in the clinical manifestations of asthma. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Monica Kraft, MD, Principal Investigator — Duke University; Dirkje S Postma, Prof. Dr., Principal Investigator — University Medical Center Groningen
Locations (26):
- United States (4):
  - Chiesi Clinical Trial Site #0503, Denver, Colorado
  - Chiesi Clinical Trial Site #0502, Durham, North Carolina
  - Chiesi Clinical Trial Site #0504, Cleveland, Ohio
  - Chiesi Clinical Trial Site #0501, Houston, Texas
- Brazil (3):
  - Prof. Dr. Emilio Pizzichini, Florianópolis
  - Prof. Dr. Alberto Cukier, São Paulo
  - Prof. Dr. Rafael Stelmach, São Paulo
- Chiesi Clinical Trial Site #0201, Montreal, Quebec, Canada
- China (3):
  - Gao, Beijing, Beijing Municipality
  - Yuanlin Song, Shanghai, Shanghai Municipality
  - Qingling Zhang, Hangzhou
- Germany (3):
  - Chiesi Clinical Trial Site #0303, Großhansdorf
  - Chiesi Clinical Trial Site #0301, Hanover
  - Chiesi Clinical Trial Site #0302, Leipzig
- Italy (6):
  - Chiesi Clinical Trial Site #0104, Ferrara
  - Chiesi Clinical Trial Site #0101, Napoli
  - Scichilone, Palermo
  - Chetta, Parma
  - Chiesi Clinical Trial Site #0103, Pisa
  - Chiesi Clinical Trial Site #0102, Verona
- Netherlands (4):
  - Dr. M. Broeders, 's-Hertogenbosch
  - W. Boersma, Alkmaar
  - Dr. J. Vroegop, Groningen
  - Dr. M. vd Berge, Groningen
- Spain (2):
  - Chiesi Clinical Trial Site #0402, Barcelona
  - Chiesi Clinical Trial Site #0401, Lugo

REFERENCES:
- [Result] Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M; ATLANTIS study group. Exploring the relevance and extent of small airways dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med. 2019 May;7(5):402-416. doi: 10.1016/S2213-2600(19)30049-9. Epub 2019 Mar 12. PMID 30876830
- [Derived] Galant SP, Kuks PJM, Kole TM, Kraft M, Siddiqui S, Fabbri LM, Beghe B, Rabe KF, Papi A, Brightling CE, Singh D, Kocks JWH, Franzini L, Vonk JM, Kerstjens HAM, Heijink IH, Pouwels SD, Slebos DJ, van den Berge M. Assessment of the role of small airway dysfunction in relation to exacerbation risk in patients with well controlled asthma (ATLANTIS): an observational study. Lancet Respir Med. 2025 Nov;13(11):990-1000. doi: 10.1016/S2213-2600(25)00283-8. Epub 2025 Sep 29. PMID 41038213
- [Derived] Kole TM, Muiser S, Kraft M, Siddiqui S, Fabbri LM, Rabe KF, Papi A, Brightling C, Singh D, van der Molen T, Nawijn MC, Kerstjens HAM, van den Berge M. Sex differences in asthma control, lung function and exacerbations: the ATLANTIS study. BMJ Open Respir Res. 2024 Jun 19;11(1):e002316. doi: 10.1136/bmjresp-2024-002316. PMID 38901877